CLINICAL TRIAL: NCT05400512
Title: Non-invasive Neuromodulation to Enhance Targeted Cognitive Remediation in Older Adults With Depression
Brief Title: Cognitive Enhancement in Depression (The COG-D Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Principal Investigator, Sarah Szymkowicz, Research Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220283
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Aging; Depression; Cognitive Symptom
Keywords: geriatrics; aging; elderly; cognition; memory; depression; tDCS; cognitive training; cognitive remediation
MeSH Terms: conditions — Depression; Neurobehavioral Manifestations | interventions — Cognitive Training; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cognitive Training + Active Stimulation (Experimental): This arm receives cognitive training combined with active tDCS.
  Interventions: Behavioral: Cognitive Training; Device: tDCS (active stimulation)
- Cognitive Training + Sham Stimulation (Experimental): This arm receives cognitive training combined with sham tDCS.
  Interventions: Behavioral: Cognitive Training; Device: tDCS (sham stimulation)

INTERVENTIONS:
Behavioral: Cognitive Training — Computerized cognitive training targeting the underlying cerebral networks associated with depression.
Device: tDCS (active stimulation) — A Soterix Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0 milliamps (mA) direct current through two bicarbon rubber electrodes encased in saline soaked 5 cm x 7 cm sponges (8 cc of 0.9% saline solution per sponge) placed over the frontal cortices at F3 and F4 (via 10-20 system).
  Arms: Cognitive Training + Active Stimulation
Device: tDCS (sham stimulation) — Sham stimulation will be performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA of direct current stimulation at the beginning of the session. Participants habituate to the sensation of tDCS within 30-60 seconds of stimulation. This procedure provides the same sensation of tDCS without the full duration of stimulation, making it a highly effective sham procedure.
  Arms: Cognitive Training + Sham Stimulation

SUMMARY:
This study will investigate whether transcranial direct current stimulation (tDCS) enhances the effects of computerized cognitive training in older adults with recurrent depression (2 or more lifetime episodes; either current or within past 3 years).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the addition of active tDCS to computerized cognitive remediation (nCCR) enhances brain activity and cognitive functions in older adults with recurrent depression to a greater degree than nCCR with sham stimulation. The investigators will randomize 20 elderly depressed outpatients to either double-blinded active or sham bifrontal tDCS plus daily nCCR over 4-weeks. Multimodal MRI (focused on the cognitive control network; CCN) and psychiatric and neuropsychological evaluations will be obtained at baseline and following intervention completion. Long-term CCN cognitive effects will be explored 3-months post-intervention via cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ years
* Diagnosis of a current or past (within last 3 years) depressive episode (e.g., Major Depressive Disorder (MDD), Persistent Depressive Disorder (PDD)) using Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria
* In total, participants must have 2 or more lifetime depressive episodes to be considered "recurrent"
* Either stable antidepressant regimen for at least 6 weeks or no current antidepressant treatment
* Evidence of subjective cognitive complaints on the Everyday Cognition Scale (ECog)
* English fluency

Exclusion criteria:

* Other Axis I psychiatric conditions via the DSM-5, except for anxiety symptoms occurring in a depressive episode
* Acute suicidality on clinical evaluation
* Acute grief
* History of alcohol use disorder or substance use disorder in last 12 months
* Currently taking medications that would significantly interact with tDCS effects (such as sodium channel blockers or anticonvulsants)
* Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury, Parkinson's disease)
* Montreal Cognitive Assessment (MoCA) score < 23
* Primary amnestic cognitive profile (>1.5 standard deviations (SDs) below demographically-adjusted mean on National Alzheimer's Coordinating Center (NACC) memory measures in context of otherwise normal cognitive profile)
* Any physical or intellectual disability affecting ability to complete assessments
* Unstable medical illness needing urgent treatment
* MRI contraindications
* Electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) in last 2 months
* Current involvement in psychotherapy
* Current involvement in other research studies (including but not limited to: neuromodulation [TMS or tDCS] or investigational drug studies)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Change in NIH Examiner scores | From baseline to post-intervention (4-6 weeks)
  This cognitive test battery assesses a range of executive functions (working memory, inhibition, set shifting, fluency, insight, and planning). The investigators will examine its Executive Composite Score, with higher scores indicate better performance.

SECONDARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) scores) | Baseline and weekly thereafter until post-intervention (4-6 weeks)
  Clinician-rated measure of depression severity, with higher scores indicative of greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M. Szymkowicz, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT05400512/ICF_002.pdf